CLINICAL TRIAL: NCT05067855
Title: Effects of Pilates Exercises on Service Speed and Agility in Squash Players
Brief Title: Effects of Pilates Exercises in Squash Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/01020 Maryam Ishfaq
Record Dates: First submitted 2021-09-24; First posted 2021-10-05 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilates exercise program group (Experimental): The pilates exercise program group will perform five exercises
  Interventions: Other: Pilates exercise program group

INTERVENTIONS:
Other: Pilates exercise program group — Pilates exercise program group will do a warm-up for 10 minutes and then perform five exercises includes standing footwork, hundreds with knee straight, articulating bridge, rolling like a ball, plank for 25 minutes. For first three weeks, each player will do 8 repetitions × 3 sets of exercises and for next three weeks, each player will do 15 repetitions × 3 sets of exercises. There will be cool-down for 10 minutes after exercises. Total program will be of 45 minutes.

SUMMARY:
To determine the effectiveness of Pilates Exercises on service speed and agility in Squash Players

DETAILED DESCRIPTION:
Squash was originated in England in the early 19th, when a group of schoolchildren noticed that punctured balls could be "squashed" against walls in a wider range of shots and it requires more effort from the player. This variation gained popularity, and the first squash courts were made in 1864; and the sport of squash was formally formed. Squash is a racquet sport in which two players compete with a hollow rubber ball on a court surrounded on four sides by walls. The players alternate hitting the ball using racquets. The ball can bounce once on the ground and as many times as the court walls allow. Squash players' main approach is to compel their opponents to go around the entire playing field. If this tactics is successful, the challenger travels a greater distance and puts a higher load on the body.

The purpose of this study is to determine the effectiveness of pilates exercises on service speed and agility in squash players.

ELIGIBILITY:
Inclusion Criteria:

* Active squash player
* Players playing squash for > 1 year
* Players engaging in squash ≥ 3 days in a week

Exclusion Criteria:

* History of any injury in past 6 months
* Those players having musculoskeletal, neurological and cardiovascular problems
* Those players who have any medical conditions

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Speed Measuring Gun | Six weeks
  Bushnell Speed Radar will be used. It uses digital technology to provide instantaneous speed measurement to +/_ .one mile per hour (MPH)/+/_.two kilometer per hour (KPH) accuracy.The Bushnell Speed Radar is a simple, point and shoot radar gun for all kinds of sports enthusiasts. The Bushnell Speed Radar measures the speed of a baseball at 10-110 MPH(16-177 KPH) from 90 feet (27 meter) away from the ball, and the speed of a racecar from 10-200 MPH (16-322 KPH) at 1,500 feet (457 meter) away. There will be two assessments, at baseline before the start of exercise program and at the end of six weeks intervention.
Badcamp Agility Test | Six weeks
  The Badcamp Agility test was performed with players standing at the middle of the badminton court. Six targets were placed at six ends of the court. The players were give warning signal and the examiner started marking the corners which players have to follow. The players have to touch all 6 markers as marked by the examiner in an undecided manner. Each participant performed the test 3 times, and the shortest time was considered for analysis. At least 1 minute of rest was given between trials. There will be two assessments, at baseline before the start of exercise program and at the end of six weeks intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Aadil Omer, Ph.D.*, Principal Investigator — Riphah International University
Locations (1):
- Sport Complex, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No